CLINICAL TRIAL: NCT04492748
Title: Collagen and PRP in Partial Thickness Rotator Cuff Injuries: Friends or Only Indifferent Neighbors: Randomized Controlled Trial
Brief Title: Rotator Cuff Tendinopathy Conservative Treatment With Collagen, PRP or Both
Acronym: RCCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sutherland Medical Center (Other)
Responsible Party: Principal Investigator, Piotr Godek, Principal Investigator, Sutherland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC2020001
Record Dates: First submitted 2020-07-20; First posted 2020-07-30 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Rotator Cuff Tendinosis; Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Collagen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collagen and PRP injections (Experimental): Ultrasound guided injections
  Interventions: Combination Product: Collagen and platelet rich plasma (PRP)
- Collagen injections (Active Comparator): Ultrasound guided injections
  Interventions: Combination Product: Collagen
- PRP injections (Active Comparator): Ultrasound guided injections
  Interventions: Combination Product: Platelet rich plasma (PRP)

INTERVENTIONS:
Combination Product: Collagen and platelet rich plasma (PRP) — Ultrasound guided injections
  Arms: Collagen and PRP injections
Combination Product: Collagen — Ultrasound guided injections
  Arms: Collagen injections
Combination Product: Platelet rich plasma (PRP) — Ultrasound guided injections
  Arms: PRP injections

SUMMARY:
The aim of the trial is comparison of the effectiveness of three methods of conservative treatment in partial thickness rotator cuff injury (PTRCI): collagen with PRP injections, PRP injections alone and collagen injections alone.

DETAILED DESCRIPTION:
BACKGROUND: Rotator cuff injury (RCI) occupy third place in the population among the musculoskeletal system pathologies (16%) after low back pain (25%) and knee pain (19%). Partial thickness RCI (PTRCI) is the sum of degenerative, overload and microtrauma processes and their incidence increases significantly with age (up to 30% over 60). One of the factors contributing to the injury is a negative collagen balance and slowed tendon metabolism in proportion to its blood supply disorders. Conservative treatment of PTRCI of degenerative origin is the first choice management, but there are no clear guidelines. External supply of collagen and PRP could potentially counteract these processes.

AIM: Comparison of the effectiveness of three treatment concepts: collagen with PRP, PRP alone, collagen alone in the treatment of PTRCI.

DESIGN: Randomized prospective trial without blinding SETTING: Open study for outpatients, single center study POPULATION: local population METHODS: Three groups of patients (each group 30 patients) with PTRCI confirmed by ultrasound (N=90). The assessment of the supraspinatus tendon (SSP) in standard position of internal rotation of the upper limb for ultrasound examination, assessment of the thickness of the RC in cross-section (mm). Each group treated by three ultrasound guided injections into the shoulder bursa every consecutive week: Group A - collagen (3 amp Collagen MD Shoulder) together with PRP (2ml); Group B - collagen alone (3 amp Collagen MD Shoulder); Group C - PRP alone. All patients were allowed to continue rehabilitation protocol. Primary control tools: NRS, QuickDash, EQ-5D-5L in control points: IA (initial assessment), 6, 12 and 24 weeks after last injection. Secondary control tools: percentage of patients where the RC continuity were preserved and percentage of patients who had ultrasonographic signs of RC regeneration (crossection width increase, improvement of echogenicity) during the observation period between W0 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs and symptoms of rotator cuff pathology
* an adult person consenting to injections
* partial thickness rotator cuff injury confirmed by ultrasound examination without coexisting severe pathologies (systemic inflammatory disease, malignancy, severe stage OA)
* no traumatic event
* no injections or any other local treatment in previous 1 month

Exclusion Criteria:

* full thickness rotator cuff injury
* acute, traumatic injuries requiring surgical treatment
* coexisting injuries of the shoulder joint requiring other intervention
* severe pathologies of the shoulder of another origin (systemic inflammatory disease, malignancy, severe stage OA)
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in EQ-5D-5L index from baseline to 24 week | Change from baseline to 24 weeks
  EQ-5D-5L index estimated from EQ-5D-5L desrcriptive system based on Polish directly measured value set. Mininmum: -0.590; Maximum: 1.0; More points means better outcome.
QuickDASH (Disabilities of Arm, Shoulder and Hand) questionnaire summary score change from baseline to 24 weeks | Change from baseline to 24 weeks
  Range: 0 (the best outcome) - 100 (the worst outcome).

SECONDARY OUTCOMES:
Pain according to Numeric Rating Scale (NRS) | Change from baseline to 6 weeks
  0 (no pain) - 10 points (the worst possible pain)
Pain according to Numeric Rating Scale (NRS) | Change from baseline to 12 weeks
  0 (no pain) - 10 points (the worst possible pain)
Pain according to Numeric Rating Scale (NRS) | Change from baseline to 24 weeks
  0 (no pain) - 10 points (the worst possible pain)
Width of rotator cuff in ultrasound imaging | Change from baseline to 24 weeks
  Dimensions of cross-section rotator cuff measure in milimeters.
Preservation of rotator cuff continuity in ultrasound imaging | Change from baseline to 24 weeks
  Presence / Absence
Regenaration of rotator cuff in ultrasound imaging | 24 weeks
  Presence / Absence
Change in EQ-5D-5L index from baseline to 6 week | Change from baseline to 6 weeks
  EQ-5D-5L index estimated from EQ-5D-5L desrcriptive system based on Polish directly measured value set. Mininmum: -0.590; Maximum: 1.0; More points means better outcome.
Change in EQ-5D-5L index from baseline to 12 week | Change from baseline to 12 weeks
  EQ-5D-5L index estimated from EQ-5D-5L desrcriptive system based on Polish directly measured value set. Mininmum: -0.590; Maximum: 1.0; More points means better outcome.
QuickDASH (Disabilities of Arm, Shoulder and Hand) questionnaire summary score change from baseline to 6 weeks | Change from baseline to 6 weeks
  Range: 0 (the best outcome) - 100 (the worst outcome).
QuickDASH (Disabilities of Arm, Shoulder and Hand) questionnaire summary score change from baseline to 12 weeks | Change from baseline to 12 weeks
  Range: 0 (the best outcome) - 100 (the worst outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Godek, PhD, Principal Investigator — Sutherland Medical Center
Locations (1):
- Sutherland Medical Center, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Godek P, Szczepanowska-Wolowiec B, Golicki D. Collagen and platelet-rich plasma in partial-thickness rotator cuff injuries. Friends or only indifferent neighbours? Randomised controlled trial. BMC Musculoskelet Disord. 2022 Dec 20;23(1):1109. doi: 10.1186/s12891-022-06089-9. PMID 36536333